CLINICAL TRIAL: NCT04740762
Title: The Effectiveness of an Individual Counselling Program in Coping With Fear of Childbirth: A Randomized Controlled Study
Brief Title: The Effect of Individual Counselling Program on Fear of Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Gizem Öztürk, Research Assistant, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Interventional study
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Fear of Childbirth; Pregnancy Related
Keywords: Prenatal care; Fear; Childbirth; Counseling; Midwifery

STUDY DESIGN:
Intervention Model Description: Following recruitment, the pregnant women were divided into a study and a control group by randomization (1:1 randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The study group were provided with individual counseling program and followed in this study, in addition to the usual care provided by healthcare professionals.
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): The control group continued to receive the routine care

INTERVENTIONS:
Behavioral: Intervention group — The women in the intervention groups were administered a three-session intervention program in addition to the routine care they received.The program encompassed providing the women with an educational booklet, childbirth stories and childbirth videos that were created to reduce their fears of childbirth.The interviews were held a total of three times, in gestational weeks 28-30, 31-33 and 34-36. The duration of the intervention at each visit was 60-80 minutes. Depending on the woman's own preference, she was invited to visit the delivery room at the second or last session and meet the midwives there. The women who did not wish to go to the delivery room were alternatively provided with photographs of the delivery room so they could take a look. Again as part of the education program, the women were given the links to the selected childbirth videos and given the opportunity to watch them.
  Arms: Intervention group

SUMMARY:
A randomized control trial was made to developing an individual counseling program to help women cope with their fear of childbirth and testing the program for effectiveness.

DETAILED DESCRIPTION:
Fear of childbirth is a common problem among women and one that affects their health and welfare before and during pregnancy and in the postpartum period. The problem can lead to adverse pregnancy outcomes and also cause a woman to experience psychological issues. Fear of childbirth can also influence the determination of the mode of delivery and can amount to a rise in cesarean rates.

The healthcare provided by midwives and other healthcare professionals during pregnancy and childbirth have the power to reduce or exacerbate childbirth fears. The most significant midwifery intervention that can be used to diminish the fear of childbirth is counseling. There is a need to develop and test individual counseling models that require the basic training skills that midwives can use as part of their routine care to address women's fears and expectations about childbirth. The individual counseling program developed in this context may be an easy-to-implement and cost-effective method to use.

This study was conducted for the purposes of developing an individual counseling program to help women cope with their fear of childbirth and testing the program for effectiveness.

It was tested the hypotheses that there is no difference between the intervention and control groups of pregnant women after the intervention in terms of fear of childbirth, childbirth self-efficacy and state anxiety scores and childbirth outcomes (duration of labor, mode of delivery, elective and emergency cesarean rates, postpartum hypertension and need for a blood transfusion, the admittance of the newborn into the intensive care unit, preferences for future births and duration of stay in hospital).

ELIGIBILITY:
Inclusion Criteria:

* Primiparas
* Ages between 18-35
* Lived in Aydın
* In gestational week 28-30,
* Pregnant with a single child
* Minimum a primary school graduate (since the questionnaires would be filled out by self-reporting)
* In a low-risk pregnancy (on the basis of the criteria of the Ministry of Health),
* Willing to divulge their own or their husband's telephone numbers,

Exclusion Criteria:

* High-risk pregnancy who had psychological and mental health problems
* History of infertility
* Speech and hearing disabilities
* Substance or narcotics users

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 70 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Fear of childbirth before intervention | 28-30 gestational weeks
  assessed using the Wijma Delivery Expectancy/Experience Questionnaire- Version A. This instrument contains questions on women's prenatal expectations to measure the nature of the fear experienced during and following childbirth. The instrument makes it possible to identify the nature of the fear of childbirth women feel before their delivery. This scale contain 33 questions. Wijma Delivery Expectancy/Experience Questionnaire- Version A is based on a 6-point Likert scale numbered 0-5. Zero corresponds to the response, "Totally" and five means "none." The minimum possible score on the scale is a "0"; maximum is 165. Higher scores indicate greater levels of Fear of Childbirth.
Fear of childbirth after intervention | 36-38 gestational weeks
  assessed using the Wijma Delivery Expectancy/Experience Questionnaire- Version A. This instrument contains questions on women's prenatal expectations to measure the nature of the fear experienced during and following childbirth. The instrument makes it possible to identify the nature of the fear of childbirth women feel before their delivery. This scale contain 33 questions. Wijma Delivery Expectancy/Experience Questionnaire- Version A is based on a 6-point Likert scale numbered 0-5. Zero corresponds to the response, "Totally" and five means "none." The minimum possible score on the scale is a "0"; maximum is 165. Higher scores indicate greater levels of Fear of Childbirth.
Fear of childbirth after birth | 12th-24th hour after the birth
  assessed using the Wijma Delivery Expectancy/Experience Questionnaire- Version B. This instrument contains questions on women's postpartum experiences to measure the nature of the fear experienced during and following childbirth. The instrument makes it possible to identify the nature of the fear of childbirth women feel after their delivery. This scale contain 33 questions. Wijma Delivery Expectancy/Experience Questionnaire- Version-B is based on a 6-point Likert scale where the responses are numbered from 1-6 and one corresponds to the response, "Totally" and six means "none." The total possible score on the scale varies between 33-198. Higher scores indicate greater levels of Fear of Childbirth.
Childbirth Self-Efficacy before intervention | 28-30 gestational weeks
  assessed using the Childbirth Self-efficacy Inventory-Short Form. The instrument measure levels of self-efficacy during labor. The scale is comprised of two subscales-outcome expectancies and self-efficacy expectancies. In the outcome expectancies subscale, responses range from 1: "not at all helpful" to 10: "very helpful," while in the self-efficacy expectancies subscale, the first 13 items are marked as 1: "Completely sure," to 10: "Not at all sure" and items 14-16 receive a score of 1: "Not at all sure" to 10: "Completely sure." All the responses to the inventory are based on a 10-point Likert-type scale. The lowest possible score on the Childbirth Self-efficacy Inventory is 32; the highest is 320. The higher the score, the more self-efficacy and confidence the pregnant woman has.
Childbirth Self-Efficacy after intervention | 36-38 gestational weeks
  assessed using the Childbirth Self-efficacy Inventory-Short Form. The instrument measure levels of self-efficacy during labor. The scale is comprised of two subscales-outcome expectancies and self-efficacy expectancies. In the outcome expectancies subscale, responses range from 1: "not at all helpful" to 10: "very helpful," while in the self-efficacy expectancies subscale, the first 13 items are marked as 1: "Completely sure," to 10: "Not at all sure" and items 14-16 receive a score of 1: "Not at all sure" to 10: "Completely sure." All the responses to the inventory are based on a 10-point Likert-type scale. The lowest possible score on the Childbirth Self-efficacy Inventory is 32; the highest is 320. The higher the score, the more self-efficacy and confidence the pregnant woman has.
State Anxiety before intervention | 28-30 gestational weeks
  assessed using the State Anxiety Inventory. The instrument is composed of 20 items. The total possible score on the instrument varies between 20-80. The measurements according to the State Anxiety Inventory scores indicate no anxiety at a score of 0-19, moderate anxiety at 20-39, a high level of anxiety at 40-59, severe anxiety at 60-79 and panic-evoking anxiety at 80 and above.
State Anxiety after intervention | 36-38 gestational weeks
  assessed using the Childbirth Self-efficacy Inventory-Short Form. The instrument measure levels of self-efficacy during labor. The scale is comprised of two subscales-outcome expectancies and self-efficacy expectancies. In the outcome expectancies subscale, responses range from 1: "not at all helpful" to 10: "very helpful," while in the self-efficacy expectancies subscale, the first 13 items are marked as 1: "Completely sure," to 10: "Not at all sure" and items 14-16 receive a score of 1: "Not at all sure" to 10: "Completely sure." All the responses to the inventory are based on a 10-point Likert-type scale. The lowest possible score on the Childbirth Self-efficacy Inventory is 32; the highest is 320. The higher the score, the more self-efficacy and confidence the pregnant woman has.
Duration of labor | 12th-24th hour after the birth
  used to determine the duration of labor. Duration of labor was recorded by the researcher to postpartum questionnaire as hours from hospital record.
Mode of Delivery | 12th-24th hour after the birth
  used to determine the mode of delivery. Mode of delivery was recorded by the researcher to the postpartum questionnaire as vaginal or cesarean section.
Elective and Emergency Cesarean Rates | 12th-24th hour after the birth
  used to determine the elective and emergency cesarean rates. Elective and emergency cesarean rates were recorded by the researcher to postpartum questionnaires as yes or no from hospital record.

SECONDARY OUTCOMES:
Postpartum hypertension | 12th-24th hour after the birth
  used to determine postpartum hypertension. Postpartum hypertension was recorded by the researcher to postpartum questionnaires as yes or no from hospital record.
Need for a blood transfusion | 12th-24th hour after the birth
  used to determine needing for a blood transfusion. Needing for a blood transfusion was recorded by the researcher from hospital record to postpartum questionnaires as yes or no depending on whether there was a blood transfusion.
Admittance of the Newborn into the Intensive Care Unit | 12th-24th hour after the birth
  used to determine the admittance of the newborn into the intensive care unit. Admittance of the Newborn into the Intensive Care Unit was recorded by the researcher from hospital records to postpartum questionnaires as yes or no depending on whether the baby was in intensive care.
Preferences for Future Births | 12th-24th hour after the birth
  used to determine the preferences for future births. Preferences for future births was measured and recorded by the researcher to postpartum questionnaires as vaginal or cesarean section.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Öztürk, PhD, Study Chair — Adnan Menderes University, Faculty of Health Sciences, Division of Midwifery
Locations (1):
- Turkey, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.